CLINICAL TRIAL: NCT04955912
Title: Effects of Music Medicine on Premenstrual Symptoms Levels and Quality of Life: A Randomized Controlled Trial
Brief Title: Music and Premenstrual Symptoms and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırklareli University (Other)
Responsible Party: Principal Investigator, Ayca Solt Kirca, Assistant Professor, Kırklareli University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KırklareliAS-3
Record Dates: First submitted 2021-06-13; First posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: MUSIC THERAPY; Premenstrual Syndrome
Keywords: Premenstrual syndrome; music medicine; quality life; midwife; nurse
MeSH Terms: conditions — Premenstrual Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Music medicine
  Interventions: Other: music medicine
- Control group (No Intervention): not routinely do anything to reduce premenstrual symptoms

INTERVENTIONS:
Other: music medicine — To reduce premenstrual symptoms by applying music medicine to people with premenstrual syndrome
  Arms: Experimental group

SUMMARY:
Premenstrual syndrome is an important health problem affecting women of childbearing age. This study is a prospective, single-blinded randomized controlled trial. Participants were randomized into music, and control groups. Immediately post-intervention, the women in the experimental groups had significantly higher reduce premenstraul syndrome levels and increase a quality life.

DETAILED DESCRIPTION:
Premenstrual syndrome is an important health problem affecting women of childbearing age. This study aimed to show that music medicine can be used to reduce premenstrual syndrome levels and increase quality of life. This study is A prospective, single-blinded randomized controlled trial. The study was conducted between January and April 2021 with 97 women who are college students. Participants consisted of women over 20 years of age and with have premenstraul snydrome. Participants were randomized into music, and control groups. Immediately post-intervention, the women in the experimental groups had a significantly higher reduce premenstraul syndrome levels and increase a quality life. Each method (music and control group) is evaluated for The Premenstrual Syndrome Scale and Short form of the WHOQOL-BREF.

ELIGIBILITY:
Inclusion Criteria:

* being between the ages of 18 and 30
* being able to speak and understand Turkish,
* having obtained a score of 45 and above from the PMSS,
* having regular menstruation (between 21-35 days),
* completing the scale forms completely and reading and approving the voluntary consent form

Exclusion Criteria:

* Having any gynecological disease (abnormal uterine bleeding, myoma, ovarian cysts, hormonal treatment, etc.),
* having a chronic or physical disease (serious hearing and vision problems, vestibular disorders that may cause balance losses),
* having any problem that prevents the person from communicating (not being able to speak Turkish, having speaking disabilities, impaired hearing, understanding abilities),
* undergoing a psychiatric treatment (pharmacotherapy or psychotherapy),
* performing one of the pharmacological or non-pharmacological practices aimed at reducing the symptoms of premenstrual symptoms (oral contraceptive use, acupressure, homeopathy, acupuncture) and exercising regularly.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 89 (Actual)
Dates: Start 2021-01-30 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Symptoms of premenstrual syndrome to reduce (PMSS) with music therapy | 14 days before application
  The female students who met the inclusion criteria were included in the study. They were randomly assigned to the music (Group 1) and control (Group 2) groups. Before starting the application, participants were asked to fill out, the The Premenstrual Syndrome Scale (PMSS). Music group: The students listened to the playlists created specifically for each participant by an expert researcher who had received music therapy training after determining the music genres they liked during a menstrual cycle (14 days before the start of the cycle) 3 times a week for 30 minutes each time.
Quality of life increase with music therapy | 14 days before application
  The female students who met the inclusion criteria were included in the study. They were randomly assigned to the music (Group 1) and control (Group 2) groups. Before starting the application, participants were asked to fill out, the The Short form of the WHOQOL-BREF (the WHOQOL-BREF). Music group: The students listened to the playlists created specifically for each participant by an expert researcher who had received music therapy training after determining the music genres they liked during a menstrual cycle (14 days before the start of the cycle) 3 times a week for 30 minutes each time.
Symptoms of premenstrual syndrome to reduce (PMSS) | 3 months
  The participants who did not state their music preference were played classical music, a music genre expected to be effective in reducing their pain and anxiety. Since the control group consisted of people who did not make any application to reduce PMSS, no application was made to this. After the application, the experimental and control groups filled with the PMSS again.
Quality of life increase | 3 months
  The participants who did not state their music preference were played classical music, a music genre expected to be effective in reducing their pain and anxiety. Since the control group consisted of people who did not make any application to reduce PMSS, no application was made to this. After the application, the experimental and control groups filled with the WHOQOL-BREF again.
The Student Information Form | 1 month
  This form consists of 25 items questioning the woman's socio-demographic characteristics (age, height, weight, living region, family type, income status), information about her menstrual cycle, duration of her first menstruation, her age at the first menstruation (menarche), presence of chronic disease, menstrual symptoms, presence of a gynecologic disease, exercise status, and music preferences
The Premenstrual Syndrome Scale (PMSS) | 3 months
  The PMSS was developed by Gençdoğan et al. (2006) to asses premenstrual symptom complaints (Gençdoğan et al., 2006). The scale is a 5-point Likert type and it consists of 44 items.The scale has nine subscales including depressive affection, anxiety, fatigue, irritability, depressive thoughts, pain, changes in appetite, sleep changes, and swelling. The premenstrual syndrome scale is administered by evaluating retrospectively, in other words, the week before the menstruation is taken into account. The overall premenstrual syndrome scale score is the sum of the scores of the nine subscales.The minimum and maximum possible scores to be obtained from this easily self-administered PMSS are 44 and 220 respectively. While the score of 44 points means no PMS, points between 45 and 103 indicate mild PMS, points between 104 and 163 indicate moderate PMS, and points between 164 and 220 severe PMS (Gençdoğan et al., 2006).
Short form of the WHOQOL-BREF | 3 months
  The World Health Organization (WHO) developed the WHOQOL-100 scale (Whoqol et al., 1998). The validity and reliability study of the Turkish version of the WHOQOL-BREF was performed by Eser (Eser et al., 1998). The WHOQOL-BREF consists of four domains, namely physical health, psychological health, social relationships, and environment. Responses given to the items are rated on a 5-point Likert type scale. The questions are answered by considering the last 15 days. The WHOQOL-BREF doesn't have a total score. The score of each domain indicates the level of quality of life for that domain. The higher the score is the better the quality of life is. The first two questions of the scale are not included in the scoring and are evaluated separately. The 3rd, 4th, and 26th questions in the scale are negatively keyed expressions (Whoqol et al., 1998; Skevington et al., 2004). While the original scale has 26 items, the Turkish version has 27 items.

CONTACTS AND LOCATIONS:
Overall Officials: AYCA SOLT KIRCA, Phd, Study Director — Kırklareli University
Locations (1):
- Kırklareli University, Kırklareli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No